CLINICAL TRIAL: NCT02253680
Title: A Prospective, Randomised Control Trial Investigating the Use of a Two-layer, Short-stretch Compression Bandage in Elective Total Knee Replacement - Feasibility
Brief Title: The Use of Compression Bandages in Total Knee Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mike Reed, Consultant Trauma and Orthopaedic Surgeon, Northumbria Healthcare NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCTTKR-01
Record Dates: First submitted 2013-09-01; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Total knee replacement; Enhanced recovery; Compression bandages
MeSH Terms: conditions — Osteoarthritis | interventions — Compression Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine care (No Intervention): Wool and crepe bandage for 24 hours post-operatively
- Compression bandage (Experimental): Actico, inelastic, short-stretch compression bandage worn 24 hours post-operatively
  Interventions: Procedure: Actico, short-stretch, inelastic dressing

INTERVENTIONS:
Procedure: Actico, short-stretch, inelastic dressing — Worn 24hr post-operatively
  Other Names: Compression bandage
  Arms: Compression bandage

SUMMARY:
The use of compression bandages in elective orthopaedic knee surgery is well regarded, however, there is a lack of robust, well-designed evidence to support this.

The aim is to determine the feasibility of conducting a randomised control trial comparing the use of a compression bandage worn post-operatively for 24 hours after elective total knee replacement, compared to standard practice (wool and crepe, non-compressive dressing).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Able to give written, informed consent
* Primary total knee replacement

Exclusion Criteria:

* Extensive peripheral vascular disease
* Lower limb neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 6 months
  Additionally, the study is a feasibility study to estimate (via the pilot trial) rates of patient recruitment, randomisation, retention and response, logistics of trial methodology, and resource utilisation.

SECONDARY OUTCOMES:
Knee range of motion | 6 months
  Range of motion of the knee compared to the pre-operative knee.
Pain | 6 months
  Post-operative pain scores measured by visual analogue scale
Patient satisfaction | 6 months
  Oxford knee score and EQ-5D scores pre-operatively and at six months

OTHER OUTCOMES:
Knee ROM | 6 months
  Circumference of knee 10cm above, at and below patella

CONTACTS AND LOCATIONS:
Overall Officials: Mike Reed, MD FRCS, Principal Investigator — Northumbria NHS Trust
Locations (2):
- United Kingdom (2):
  - Wansbeck District General Hospital, Ashington, Northumberland
  - Northumbria Healthcare NHS Foundation Trust, Ashington